CLINICAL TRIAL: NCT04979897
Title: Impact on Mental, Physical, And Cognitive Functioning of a Critical Care sTay During the COVID-19 Pandemic (IMPACCT COVID-19): a Prospective, Multicentre, Mixed-methods Cohort Study
Brief Title: Impact on Mental, Physical, And Cognitive Functioning of a Critical Care sTay During the COVID-19 Pandemic
Acronym: IMPACCT
Status: Completed | Type: Observational
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Clinica Alemana de Santiago (Other); Clinica Indisa (Other); Clinica Bupa Santiago (Other); Hospital del Salvador (Other); Hospital Clínico Regional De Antofagasta Dr Leonardo Guzman (Other); Hospital San Pablo de Coquimbo (Other); Hospital Metropolitano (Other)
Responsible Party: Principal Investigator, Ana Cristina Castro, Visiting lecturer, Universidad del Desarrollo
Other Study IDs: 2020-78
Record Dates: First submitted 2021-07-24; First posted 2021-07-28 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Covid19; Critical Care; Postintensive Care Syndrome
Keywords: Covid19; Critical care; Postintensive Care Syndrome; Rehabilitation; Follow-up
MeSH Terms: conditions — COVID-19; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive care unit stay during high bed occupancy in the COVID-19 pandemic: Adult patients (≥18 years old) who are mechanically ventilated for at least 48 hours in one of the participating ICUs during a high bed occupancy in the pandemic
  Interventions: Other: Intensive care unit stay during the COVID-19 pandemic
- Intensive care unit stay during low bed occupancy in the COVID-19 pandemic: Adult patients (≥18 years old) who are mechanically ventilated for at least 48 hours in one of the participating ICUs during a low bed occupancy in the pandemic
  Interventions: Other: Intensive care unit stay during the COVID-19 pandemic

INTERVENTIONS:
Other: Intensive care unit stay during the COVID-19 pandemic — Patients will be screened daily for a potential ICU discharge. Each site coordinator, which is a clinician physiotherapist responsible for the site, will check that the patient is delirium-free (CAM-ICU negative) and cooperative (i.e. using 5 standardised questions: open [close] your eyes; look at me; open your mouth and stick out your tongue; nod your head; raise your eyebrows when I have counted up to five) within 72 hours from ICU discharge. Every patient deemed eligible will be invited to participate through a face-to-face visit by the assigned evaluator, receiving verbal and written information about the study

SUMMARY:
Intensive care unit (ICU) survivors and their families frequently present mental, cognitive and physical impairments lasting years. The ongoing pandemic could affect the duration, variety, and severity of these impairments. Our aim is to determine the impact of the COVID-19 pandemic on the physical, mental, and cognitive health of survivors, the experience of their families and their treating healthcare professionals in the long-term.

This is a prospective, multicentre, mixed-methods cohort study in seven Chilean ICUs. The perceptions of family members regarding the ICU stay and the later recovery will be explored 3 months after discharge. Health care professionals will be invited to discuss the challenges faced during the pandemic using semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Mechanically ventilated for at least 48 hours

Exclusion Criteria:

* Unable to walk independently 2 weeks prior to ICU admission (with or without a gait aid)
* S5q < 5 or CAM-ICU positive within 72 hours after ICU discharge
* Patient who do not understand or speak Spanish
* Patient unable to communicate verbally
* Burn or severe trauma as admission diagnosis
* Any neurological disorder (i.e. spinal cord injury, stroke and brain tumours) as admission diagnosis
* Transferred to a non-participating study centre before ICU discharge assessment
* Recent prolonged hospital stay (extended by more than 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who were mechanically ventilated in the ICU, either with the diagnosis of COVID-19 or other causes
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Castro-Ávila, PhD, Principal Investigator — Universidad del Desarrollo
Locations (7):
- Chile (7):
  - Hospital Regional Dr. Leonardo Guzmán de Antofagasta, Antofagasta
  - Hospital San Pablo de Coquimbo, Coquimbo
  - Clínica Alemana de Santiago, Santiago
  - Clínica BUPA, Santiago
  - Clínica INDISA, Santiago
  - Hospital del Salvador, Santiago
  - Hospital Metropolitano, Santiago

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Castro-Avila A, Merino-Osorio C, Gonzalez-Seguel F, Camus-Molina A, Munoz-Munoz F, Leppe J; IMPACCT COVID-19 study group. Six-month post-intensive care outcomes during high and low bed occupancy due to the COVID-19 pandemic: A multicenter prospective cohort study. PLoS One. 2023 Nov 16;18(11):e0294631. doi: 10.1371/journal.pone.0294631. eCollection 2023. PMID 37972091
- [Derived] Castro-Avila AC, Merino-Osorio C, Gonzalez-Seguel F, Camus-Molina A, Leppe J; IMPACCT COVID-19 study group. Impact on Mental, Physical and Cognitive functioning of a Critical care sTay during the COVID-19 pandemic (IMPACCT COVID-19): protocol for a prospective, multicentre, mixed-methods cohort study. BMJ Open. 2021 Sep 8;11(9):e053610. doi: 10.1136/bmjopen-2021-053610. PMID 34497087
- See also: Custom-made study web site — https://medicina.udd.cl/kinesiologia-santiago/impacct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 20th, 2020 to April 12th, 2021
Pre-assignment Details: Not recruited (n=152)
  * Declined to participate (n=18)
  * Unable to cooperate (n=40)
  * Lack of evaluator (n=94)
Period: Overall Study
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Started | 149 | 103
3-month Follow-up | 55 | 50
Completed | 30 | 37
Not Completed | 119 | 66
Not completed — Death | 1 | 8
Not completed — Lost to Follow-up | 111 | 56
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic | Total
Number analyzed (Participants) | 149 | 103 | 252
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [44 to 63] | 61 [51 to 71] | 57 [47 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 41 | 89
  Male | 101 | 62 | 163
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: The WHODAS 2.0 is a self-reported disability questionnaire based on the International Classification of Functioning, Disability, and Health (ICF). It includes 36 questions, organised under six domains (cognition, mobility, self-care, getting along, life activities and participation). Each question must be answered based on the perceived difficulty for performing activities using a 5-point scale (none, mild, moderate, severe and extreme). The overall score of each domain, it is transformed into a score between 0 and 100, where 0 means no disability and 100 is complete disability
Time Frame: 6 months after the ICU discharge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 30 | 37
units on a scale | 5 [2 to 18] | 13.5 [2 to 23]

2. Secondary Outcome: Clinical Frailty Scale
Description: The CFS evaluates specific domains including physical functioning, activities of daily living (ADL), instrumental ADL, assistance for personal care, comorbidities, and cognition to generate a frailty score using a 9-point scale ranging from 1 (very fit) to 9 (terminally ill). A score greater than 4 is considered fragile
Time Frame: Within 72 hours from ICU discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 149 | 103
score on a scale | 2 [2 to 3] | 3 [2 to 3]

3. Secondary Outcome: Medical Research Council Sum Score (MRC-SS): Peripheral Muscle Strength
Description: the MRC-SS consists of a standardised examination of six muscle groups bilaterally (i.e. shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension and dorsiflexion). All muscle groups are scored using a 6-point scale between 0 and 5 (0 = no visible /palpable contraction; 1 = visible / palpable contraction or no limb movement; 2 = limb movement, but not against gravity; 3 = movement against the gravity over nearly the entire range of motion; 4 = motion against gravity and resistance, subjectively adjusted for gender and age; 5 = normal force). The score goes from 0 (no strength) to a maximum score of 60 points, indicating normal peripheral strength.
Time Frame: Within 72 hours from ICU discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 149 | 103
score on a scale | 52 [46 to 57] | 50 [44 to 57]

4. Secondary Outcome: Functional Status Score for the Intensive Care Unit (FSS-ICU)
Description: The FSS-ICU is a mobility instrument to score the level of physical assistance required when performing five functional activities: rolling, transfer from supine to sit, sitting at the edge of the bed, transfer from sitting to stand, and walking. Each activity is scored using a 7-point scale ranging from 0 (not able to perform) to 7 (complete independence). The resulting overall score ranges from 0 to 35 points, where a higher scores indicates better performance.
Time Frame: Within 72 hours from ICU discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 149 | 103
score on a scale | 26 [21 to 32] | 27 [19 to 32]

5. Secondary Outcome: Montreal Cognitive Assessment-Blind (MoCA Blind)
Description: The MoCA blind is a cognitive screening tool designed to detect cognitive dysfunction in five areas: memory, attention, language, abstraction and orientation. Each domain is scored separately for a total score ranging from 0 to 22 points. A score equal to or greater than 18 points is considered normal cognition.
Time Frame: 6 months after the ICU discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 30 | 37
score on a scale | 21 [19 to 22] | 20 [18 to 22]

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is an interviewer or self-administered questionnaire designed to identify anxiety and depressive symptoms in a wide variety of in-hospital patients, which requires between 2 and 5 minutes to be completed. The HADS has fourteen questions, seven for anxiety and seven for depressive symptoms. Each question is rated with a 4-point scale ranging from 0 ("absence") to 3 ("extreme presence"), resulting in a sum score of 21 points per subscale. For each subscale, a score >8 indicates suspected anxiety or depression, while a score >11 indicates clinical symptoms of anxiety or depression.
Time Frame: 6 months after the ICU discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 30 | 37
score on a scale
  Depression subscale | 7 [5 to 8] | 7 [5 to 9]
  Anxiety subscale | 6 [3 to 9] | 7 [3 to 10]

7. Secondary Outcome: Impact of Events Scale-Revised (IES-R)
Description: The IES-R is an interviewer or self-administered questionnaire designed to measure the subjective distress caused by traumatic events that has been validated for critical illness survivors. It comprises 22 questions in three subscales: intrusion, avoidance, and hyperarousal. Questions are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The score goes from 0 to 88 points. Scores above 33 are indicative of post-traumatic stress symptoms.
Time Frame: 6 months after the ICU discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 30 | 37
score on a scale | 13.5 [5 to 38] | 22 [7 to 44]

8. Secondary Outcome: European Quality of Life Health Questionnaire (EQ-5D-3L)
Description: The EQ-5D-3L is an interviewer or self-administered questionnaire of health status or health-related quality of life, including five domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression and global health state. Each domain is scored based on 3 levels of severity: no problems, some problems, and extreme problems. Each combination of answers can be translated into a utility score, where 0 is similar to being dead and 1 represents the best possible quality of life. The utility scores were obtained using the Chilean Social valuation of EQ-5D health states (DOI: http://dx.doi.org/10.1016/j.jval.2011.09.002)
Time Frame: 6 months after the ICU discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 30 | 37
score on a scale | 0.79 [0.57 to 1.00] | 0.74 [0.51 to 0.79]

9. Secondary Outcome: Employment Status
Description: The employment status was evaluated using the following questions: What is your current employment status? What working hours do you have? and has your employment situation changed after your ICU stay?
Time Frame: 6 months after the ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 30 | 37
Participants
  Employed-Full time | 18 | 17
  Employed-Part time | 3 | 3
  Umemployed | 4 | 9
  Retired | 4 | 8
  No answer | 1 | 0

10. Secondary Outcome: Survival
Description: Number of patients who survived
Time Frame: 6 months after the ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 149 | 103
Participants | 148 | 95

11. Other Pre Specified Outcome: Cohort Retention Rate
Description: Number of patients who can be contacted and evaluated
Time Frame: Every month during one year
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
Number analyzed (Participants) | 149 | 103
Participants | 30 | 37

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intensive Care Unit Stay During High Bed Occupancy in the COVID-19 Pandemic | Intensive Care Unit Stay During Low Bed Occupancy in the COVID-19 Pandemic
All-Cause Mortality (participants affected / at risk) | 1/149 | 8/103
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/103
Other Adverse Events (participants affected / at risk) | 0/149 | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04979897/Prot_SAP_000.pdf